CLINICAL TRIAL: NCT02822846
Title: Evaluation of Diagnostic Qualities of Lung Ultrasonography to Monitor the Position of the Intubation Probe
Brief Title: Evaluation of the Ability to Diagnose the Position of the Intubation Probe Thanks to Lung Ultrasonography
Acronym: ECOVERA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-04-07
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Intubation, Intratracheal
Keywords: Lung ultrasound; Sliding lung; Probe position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: lung ultrasound

SUMMARY:
The purpose of this study is to evaluate the diagnostic qualities of lung ultrasonography to monitor the position of the intubation probe.

The primary assessment criterion is of study the position of the intubation probe with two examinations carried out independently :

* sonography
* chest radiography

A correct position of the intubation probe will be considered if there is :

* Highlighting of the extremity of the intubation probe in endo tracheal
* Highlighting bilateral lung sliding

DETAILED DESCRIPTION:
Oesophageal intubation can cause death. Selective intubation can induce a poor ventilation, hypoxemia, atelectasis etc… It's not rare in paediatric intubation. The prevalence of malposition of endotracheal tube is 30 to 40% in babies and infants less than 1 year old. Currently doctors try to detect malposition of intra-tracheal tube by auscultation and capnograms and chest radiography is needed to confirm it. The Chest X ray is the gold standard.

The aim of the study is to confirm the good positioning of the tube with a lung ultrasonography.

After each intra-tracheal intubation, for patients with qualifying criteria, a lung ultrasonography will be performed, in bed, by two trained doctors (senior and junior) to determine if the position is right. Then, the chest radiography will be performed as usual.

ELIGIBILITY:
Inclusion Criteria:

* Patient less than 18 years old
* Patient intubated and ventilated
* intubation probe considered in place on auscultation
* SpO2> 92%
* Affiliate or entitled to a social security scheme
* No opposition of any of the parents.

Exclusion Criteria:

* Children too unstable : decompensated shock
* Spontaneous pneumothorax
* Heart massage ongoing
* Chest trauma
* Faulty position of the probe intubation

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Intubated and ventilated minors
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-11-19 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the position of intubation probe by comparison between chest radiography and lung ultrasonography | day of enrollment
  correct position is defined by :
  * visualization of the probe intubation extremity in endotracheal
  * visualization of bilateral lung sliding

SECONDARY OUTCOMES:
Number of patients with malposition of the oesophageal or selective intubation probe | day of enrollment
Number of mobilized intubation probes | day of enrollment
  Due to inefficient ventilation and despite undetected malposition
Number of malpositions of the intubation probe evaluated with lung ultrasonography by junior evaluator | day of enrollment
Number of malpositions of the intubation probe evaluated with lung ultrasonography by senior evaluator | day of enrollment
Number of malpositions of the intubation probe evaluated with a chest radiography by junior evaluator | day of enrollment
Number of malpositions of the intubation probe evaluated with a chest radiography by senior evaluator | day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Julie Starck, MD, Principal Investigator — AP-HP, Necker hospital
Locations (1):
- Intensive Care Unit of Necker Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knapp S, Kofler J, Stoiser B, Thalhammer F, Burgmann H, Posch M, Hofbauer R, Stanzel M, Frass M. The assessment of four different methods to verify tracheal tube placement in the critical care setting. Anesth Analg. 1999 Apr;88(4):766-70. doi: 10.1097/00000539-199904000-00016. PMID 10195521
- [Background] Harris EA, Arheart KL, Penning DH. Endotracheal tube malposition within the pediatric population: a common event despite clinical evidence of correct placement. Can J Anaesth. 2008 Oct;55(10):685-90. doi: 10.1007/BF03017744. PMID 18835966
- [Background] Schmolzer GM, O'Reilly M, Davis PG, Cheung PY, Roehr CC. Confirmation of correct tracheal tube placement in newborn infants. Resuscitation. 2013 Jun;84(6):731-7. doi: 10.1016/j.resuscitation.2012.11.028. Epub 2012 Dec 1. PMID 23211476
- [Background] Chou EH, Dickman E, Tsou PY, Tessaro M, Tsai YM, Ma MH, Lee CC, Marshall J. Ultrasonography for confirmation of endotracheal tube placement: a systematic review and meta-analysis. Resuscitation. 2015 May;90:97-103. doi: 10.1016/j.resuscitation.2015.02.013. Epub 2015 Feb 21. PMID 25711517
- [Background] Pfeiffer P, Rudolph SS, Borglum J, Isbye DL. Temporal comparison of ultrasound vs. auscultation and capnography in verification of endotracheal tube placement. Acta Anaesthesiol Scand. 2011 Nov;55(10):1190-5. doi: 10.1111/j.1399-6576.2011.02501.x. Epub 2011 Sep 8. PMID 22092123
- [Background] American College of Emergency Physicians. Clinical Policies Committee. Verification of endotracheal tube placement. Ann Emerg Med. 2002 Nov;40(5):551-2. No abstract available. PMID 12425285
- [Background] Guerder M, Maurin O, Merckx A, Foissac F, Oualha M, Renolleau S, Vedrenne-Cloquet M. Diagnostic value of pleural ultrasound to refine endotracheal tube placement in pediatric intensive care unit. Arch Pediatr. 2021 Nov;28(8):712-717. doi: 10.1016/j.arcped.2021.09.006. Epub 2021 Oct 6. PMID 34625381